CLINICAL TRIAL: NCT07223307
Title: Phase II Trial of REal Time MRI GUided Adaptive Stereotactic Ablative Radiotherapy for Liver Cancers Using a Single Session, Simulation Free Workflow
Brief Title: REGULUS: MRI-guided Adaptive SABR for Liver Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-82587
Record Dates: First submitted 2025-10-23; First posted 2025-10-31 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Liver Cancer; Intrahepatic Cholangiocarcinoma; Liver Metastases; HCC
MeSH Terms: conditions — Liver Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MRI-guided Adaptive Stereotactic Ablative Body Radiotherapy (SABR) (Experimental): Participants will receive a single fraction of MRI-guided adaptive stereotactic ablative body radiotherapy (SABR) using the MRIdian system. Treatment includes daily adaptive planning based on MRI to optimize dose delivery to the tumor and minimize dose to surrounding normal tissue. Eovist contrast is administered before treatment to enhance visualization. Patients perform an inspiratory breath hold during radiation delivery to minimize motion.
  Interventions: Radiation: MRI-guided adaptive stereotactic ablative body radiotherapy (SABR)

INTERVENTIONS:
Radiation: MRI-guided adaptive stereotactic ablative body radiotherapy (SABR) — A single fraction of MRI-guided adaptive stereotactic ablative body radiotherapy (SABR) will be delivered using the MRIdian system. Treatment includes adaptive planning based on daily MRI imaging to update tumor and organ-at-risk contours and optimize the radiation dose. On the day of treatment, Eovist contrast is administered 20 minutes before therapy to enhance tumor visualization. Patients perform an inspiratory breath hold during radiation delivery to minimize motion. The total dose is 30-40 Gy delivered in one fraction using external beam techniques.

SUMMARY:
Single arm unblinded study of simulation-free MRI-guided SABR with adaptive replanning in one session for treatment of patients with liver cancers

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC, intrahepatic cholangiocarcinoma, or metastatic cancer. In the case of suspected HCC in patients with known cirrhosis, noninvasive criteria recommended by the European Association for the Study of Liver Diseases (lesion > 1 cm with arterial phase hyperenhancement and venous phase washout) or LI-RADS score of 5 may be used
* ≥ 18 years old at time of study enrollment
* Child-Pugh A status
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life Expectancy > 6 months
* For women of childbearing potential or who are not postmenopausal (see Appendix F for Definition of Menopausal Status), a negative urine or serum pregnancy test must be done.
* Ability to understand and the willingness to provide written informed consent.
* Patients treated with prior liver-directed therapies with the exception of radioembolization are eligible for this study if they otherwise meet eligibility criteria

Exclusion Criteria:

* Prior treatment with radioembolization
* Cytotoxic chemotherapy or investigational agent within 1 week of SABR
* Prior radiotherapy overlapping with study treatment site
* Female patients who are pregnant
* Contraindication to having an MRI scan or inability to tolerate MRI
* Presence of a pacemaker or other implanted cardiac device
* Direct tumor extension into the stomach, duodenum, small bowel or large bowel
* Patient unable to breath hold > 15 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
1-year Overall Survival (OS) | 1 year after SABR
  Overall survival will be defined as the time from treatment to death from any cause. Patients alive at the time of analysis will be censored at last follow-up.

SECONDARY OUTCOMES:
Rate of Grade ≥ 2 Gastrointestinal (GI) Adverse Events | Within 90 days of completing SABR
  Proportion of participants experiencing CTCAE v5.0 grade ≥ 2 gastrointestinal adverse events (including fatigue, nausea, diarrhea, or GI pain) attributable to SABR.
Rate of Grade ≥ 2 Radiation Pneumonitis | Within 90 days of completing SABR
  Proportion of participants experiencing CTCAE v5.0 grade ≥ 2 radiation pneumonitis attributable to SABR.
Rate of Grade ≥ 2 Chest Wall Toxicity | Within 90 days of completing SABR
  Proportion of participants experiencing CTCAE v5.0 grade ≥ 2 chest wall toxicity attributable to SABR.
Change from Baseline in EORTC QLQ-C30 Global Health Status/Quality of Life Score up to 1 Year Post-SABR | Up to 1 year post-SABR
  Patient-reported global health status and quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).
  Scores range from 0 to 100, with higher scores indicating better global health status and overall quality of life.
Change from Baseline in FACT-Hep Total Score up to 1 Year Post-SABR | Up to 1 year post-SABR
  Patient-reported quality of life will be evaluated using the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire.
  The FACT-Hep consists of the FACT-General (FACT-G) plus additional hepatobiliary-specific items.
  Total scores range from 0 to 180, with higher scores indicating better health-related quality of life.
Change from Baseline in COST-FACIT Total Score up to 1 Year Post-SABR | Up to 1 year post-SABR
  Financial toxicity will be assessed using the Comprehensive Score for Financial Toxicity (COST-FACIT) questionnaire.
  Scores range from 0 to 44, with higher scores indicating lower financial toxicity (better financial well-being).
Rate of Patients With Total Delivery Time > 120 Minutes | Baseline
  Percentage of patients with total SABR delivery time exceeding 120 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States